CLINICAL TRIAL: NCT02673554
Title: The Reduced Insulinotropic Effect of a Continuous Infusion Relative to a Bolus Injection of Glucose-dependent Insulinotropic Polypeptide (GIP) in Patients With Type 2 Diabetes is Not Caused by Rapid Tachyphylaxis
Brief Title: The Reduced Insulinotropic Effect of a Continuous Infusion Relative to a Bolus Injection of GIP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Diabeteszentrum Bad Lauterberg im Harz (Other)
Responsible Party: Principal Investigator, Michael A. Nauck, Prof. Dr. med. Michael A. Nauck, Diabeteszentrum Bad Lauterberg im Harz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GIP and Tachyphylaxis
Record Dates: First submitted 2016-01-28; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes
Keywords: Glucose-dependent Insulinotropic Polypeptide (GIP); Glucagon-Like Peptide 1 (GLP-1); Incretin; Insulin secretion; Tachyphylaxis
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oral glucose tolerance test (Experimental): An oral glucose challenge (75 g)
  Interventions: Procedure: Oral glucose tolerance test (OGTT)
- GIP Bolus (Active Comparator): Hyperglycemic clamp (capillary venous glucose concentration ~ 8.5 mmol/l) with two repeated intravenous bolus injections of synthetic human GIP (50 pmol/kg body weight) administered 30 and 120 min after commencing the hyperglycemic clamp
  Interventions: Drug: GIP Bolus; Procedure: hyperglycemic clamp
- GIP Infusion (Active Comparator): Hyperglycemic clamp with the continuous intravenous infusion of 2 pmol.kg-1.min-1 synthetic human GIP between 30 and 180 min
  Interventions: Drug: GIP Clamp; Procedure: hyperglycemic clamp

INTERVENTIONS:
Drug: GIP Bolus — bolus injections of synthetic human GIP (50 pmol/kg body weight) administered 30 and 120 min after commencing the hyperglycemic clamp
  Arms: GIP Bolus
Drug: GIP Clamp — hyperglycemic clamp with the continuous intravenous infusion of 2 pmol.kg-1.min-1 synthetic human GIP between 30 and 180 min
  Arms: GIP Infusion
Procedure: Oral glucose tolerance test (OGTT) — an oral glucose challenge (75 g)
  Arms: Oral glucose tolerance test
Procedure: hyperglycemic clamp — a hyperglycemic clamp (capillary venous glucose concentration ~ 8.5 mmol/l)
  Arms: GIP Bolus; GIP Infusion

SUMMARY:
In patients with type 2 diabetes, the incretin hormone glucose-dependent insulinotropic polypeptide (GIP) has lost its insulinotropic activity, but more so after continuous versus bolus administration. The design was a two-way crossover design comparing repeated bolus injection and continuous infusion of GIP under hyperglycaemic clamp conditions. Patients were age- gender- and weight-matched with type 2 diabetes, first degree relatives of such patients, and healthy subjects. Investigators performed a:

1. Oral glucose challenge;
2. hyperglycemic clamp (8.5 mmol/l) with two repeated GIP bolus administrations (50 pmol/kg body weight at 30 and 120 min); and
3. hyperglycemic clamp with continuous administration of GIP (2 pmol.kg-1.min-1 from 30-180 min).

To answer the question, whether rapid tachyphylaxis occurs with regard to the insulinotropic action of GIP, investigators studied type 2-diabetic patients, their first-degree relatives, and healthy controls under hyperglycaemic clamp conditions with two GIP bolus injections 90 min apart, and compared this to a continued intravenous infusion of GIP.

ELIGIBILITY:
Inclusion Criteria:

* Exclusion of pregnancy
* Exclusion of impaired glucose tolerance or type 2 diabetes in metabolical healthy subjects
* current diagnosis of type 2 diabetes according to the guidelines of the German Diabetes Association (DDG) ( Kerner et al . 2001) in subjects of diabetes group
* fasting glucose ≤ 150 mg/dl
* Body-mass-index ≥ 20 kg/m²
* Written consent

Exclusion Criteria:

* Type 1 diabetes
* Impaired glucose tolerance or Type 2 diabetes in metabolical healthy subjects
* Ketone bodies urine diagnostics at least ++
* Acidosis
* Fasting blood glucose > 150 mg/dl
* Body-mass-index < 20 kg/m²
* No written consent
* Pregnancy or unsafe contraception in women before menopause
* Active malignancy
* Angina as current, unsolved clinical problem
* Inadequately treated or untreated arterial hypertension ( > 160 mmHg systolic and / or > 95 mmHg diastolic )
* Infection / fever > 37.5 ° C
* Treatment with glucocorticoids
* Insulin therapy within the last three months
* Anemia with a hemoglobin level < 12 g/dl
* Liver function limitations
* Renal impairment ( serum creatinine > 1.5 mg/dl )
* Alcohol or drug abuse
* Participation in clinical trials in the last 3 months
* Inability or unwillingness to comply with the requirements of the Protocol
* Known hypersensitivity to GIP

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-05; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Insulin secretory response after GIP bolus or infusion. | 210 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Nauck, Prof., Principal Investigator — Diabeteszentrum Bad Lauterberg

IPD SHARING:
Plan to Share IPD: No